CLINICAL TRIAL: NCT02171624
Title: A Two-way Crossover Study to Evaluate the Safety and Pharmacokinetics of Quinidine Sulfate Alone (200 mg Orally q2h to a Maximum of 1,000 mg), Dabigatran Etexilate Alone (150 mg BID for Three Days), and the Co-administration of Dabigatran Etexilate (150 mg BID) With Quinidine Sulfate (200 mg q2h)
Brief Title: Safety and Pharmacokinetics of Quinidine Alone and in Combination With Dabigatran Etexilate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.90
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Quinidine

ARMS (2):
- dabigatran etexilate (Experimental): quinidine run-in, followed by dabigatran+quinine and dabigatran alone in randomized order
  Interventions: Drug: dabigatran etexilate; Drug: quinidine
- quinidine (Experimental): quinidine run-in, followed by dabigatran+quinine and dabigatran alone in randomized order
  Interventions: Drug: dabigatran etexilate; Drug: quinidine

INTERVENTIONS:
Drug: dabigatran etexilate
Drug: quinidine

SUMMARY:
Open-label, two-way crossover design with a quinidine sulfate run-in period followed by a randomised sequence of dabigatran etexilate plus quinidine sulfate or dabigatran etexilate alone to evaluate the safety of co-administration of dabigatran etexilate and quinidine. and the pharmacokinetic interaction between quinidine and dabigatran etexilate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects
* Age ≥18 and Age ≤55 years
* Body Mass Index (BMI) ≥18.5 and BMI <30 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion Criteria:

* Any finding of the medical examination (including Blood Pressure (BP), Pulse Rate (PR) and Electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within thirty days prior to administration or during the trial
* Inability to refrain from smoking on trial days Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Taking drugs which are known P-gp and/or CYP3A4 inhibitors or inducers (verapamil, phenothiazine antipsychotics, macrolide antibiotics (clarithromycin, erythromycin), antifungal drugs, antiviral drugs (protease inhibitors like nelfinavir) or St. John´s Wort) within the last 4 weeks before screening
* Taking drugs which are known CYP2D6 substrates (antidepressants, antiarrhythmics, beta blockers) within the last 2 weeks before screening
* For female subjects:

  * Pregnancy or planning to become pregnant within 2 months of study completion
  * Positive pregnancy test
  * No adequate contraception e.g., sterilisation, IUD (intrauterine device), have not been using a barrier method of contraception for at least 3 months prior to participation in the study
  * Are not willing or are unable to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and up to 2 months after completion/termination of the trial
  * Chronic use of oral contraception or hormone replacement containing ethinyl estradiol as the only method of contraception
  * Partner is unwilling to use condoms
  * Currently lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Differences between treatments in systolic blood pressure profiles (using area under the BP-time curve) | -0:15 before, and every 15 minutes for 2 hours post-dose, 3, 4 and 12 hours post dose
Incidence of symptomatic hypotension | -0:15 before, and every 15 minutes for 2 hours post-dose, 3, 4 and 12 hours post dose

SECONDARY OUTCOMES:
Area under the effect curve (AUEC) for activated partial thromboplastin time (aPTT), thrombin time (TT) and ecarin clotting time (ECT) | up to 48 hours after last dose
Maximum effect ratio (ERmax) for activated partial thromboplastin time (aPTT), thrombin time (TT) and ecarin clotting time (ECT) | up to 48 hours after last dose
Occurrence of Adverse Events | up to day 26
Abnormal findings in physical examination | up to day 26
Changes from baseline in Vital Signs (Blood Pressure (BP), Heart Rate (HR)) | up to day 26
Changes from baseline in 12-lead ECG (electrocardiogram) | up to day 26
Changes from baseline in QT prolongation | up to day 26
Changes in clinical laboratory tests | up to day 26
Number of patients with adverse events leading to treatment discontinuation | up to day 26
AUC (area under the concentration-time curve of the analyte in plasma) | up to 48 hours after the last dose
Cmax (maximum measured concentration of the analyte in plasma) | up to 48 hours after the last dose
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 48 hours after the last dose
λz (terminal rate constant in plasma) | up to 48 hours after the last dose
t½ (terminal half-life of the analyte in plasma) | up to 48 hours after the last dose
Cpre (pre-dose concentration of the analyte in plasma immediately before administration of the following dose) | up to 48 hours after the last dose
MRTpo,ss (mean residence time of the analyte in the body at steady state after po administration) | up to 48 hours after last dose
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following an extravascular dose) | up to 48 hours after last dose
CL/F,ss (apparent clearance of the analyte in the plasma at steady state after extravascular administration) | up to 48 hours after last dose
Cavg (average concentration of the analyte in plasma under steady-state conditions) | up to 48 hours after last dose
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state) | up to 48 hours after last dose
PTF (peak trough fluctuation) | up to 48 hours after last administration
RAUCt1-t2, MET, 5 (ratio of AUCt1-t2 of 3-OH-quinidine/quinidine) | up to 48 hours after last dose